CLINICAL TRIAL: NCT04306926
Title: A Open-label, Single-arm, Phase II Study of TQB2450 Injection Combined With Stereotactic Body Radiation Therapy (SBRT) in Subjects With Advanced Oligometastatic Non-Small Cell Lung Cancer
Brief Title: A Study of TQB2450 Injection Combined With Stereotactic Body Radiation Therapy (SBRT) in Subjects With Advanced Oligometastatic Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2450-II-05
Record Dates: First submitted 2020-03-11; First posted 2020-03-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2019-11

CONDITIONS: Advanced Oligometastatic Non-small Cell Lung Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2450+SBRT (Experimental): SBRT three days before TQB2450.
  Interventions: Drug: TQB2450; Radiation: SBRT

INTERVENTIONS:
Drug: TQB2450 — TQB2450 1200mg administered IV on Day 1 of each 21-day cycle.
Radiation: SBRT — Give according to the location of the lesion and clinical condition.

SUMMARY:
TQB2450 is a humanized monoclonal antibody targeting programmed death ligand-1 (PD-L1), which prevents PD-L1 from binding to PD-1 and B7.1 receptors on T cell surface, restores T cell activity, thus enhancing immune response and has potential to treat various types of tumors.

ELIGIBILITY:
Inclusion Criteria:

* 1. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 2; Life expectancy ≥ 3 months.

  2. Histologically or pathologically confirmed advanced non-small cell lung cancer.

  3. Primary lesion controlled oligometastatic patients, the number of metastatic lesions ≤ 5, and has at least one measurable lesion.

  4. Has received standard first-line chemotherapy, intolerable or inappropriate to the chemotherapy.

  5. Adequate organ system function. 6. Male or female subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 6 months after the last dose of study (such as intrauterine devices , contraceptives or condoms) ；No pregnant or breastfeeding women, and a negative pregnancy test are received within 7 days before the first administration.

  7.Understood and Signed an informed consent form.

Exclusion Criteria:

* 1. Has used against PD-1, PD-L1 and other related immunotherapeutic drugs. 2.Has mutations in (epidermal growth factor receptor)EGFR, (anaplastic lymphoma kinase)ALK, (c-ros oncogene 1 receptor kinase)ROS1 or T790M and not resistant to targeted drug.

  3. Has severe hypersensitivity reaction to other monoclonal antibodies. 4. Has diagnosed and/or treated additional malignancy within 5 years prior to the first administration.Exceptions include cured basal cell carcinoma of skin and carcinoma in situ of cervix.

  5. Has any active autoimmune disease or a history of autoimmune disease. 6. Immunosuppressive therapy with immunosuppressive agents or systemic or absorbable local hormones (dosage > 10 mg/day prednisone or other therapeutic hormones) is required for the purpose of immunosuppression, and is still in use for 2 weeks after the first administration.

  7. (Magnetic Resonance Imaging)MRI examination found meningeal metastases and cannot be controlled by stereotactic radiotherapy.

  8. Has adverse events caused by previous therapy except alopecia that did not recover to ≤grade 1.

  9. Has any severe and/or uncontrolled disease. 10. Has vaccinated with vaccines or attenuated vaccines within 4 weeks prior to first administration.

  11. According to the judgement of the researchers, there are other factors that may lead to the termination of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2022-10-31 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Baseline up to 96 weeks
  PFS was defined as the time from the date of study enrollment to the date of the first of the following events, objective disease progression or death due to any cause.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Baseline up to 96 weeks
  Percentage of subjects achieving complete response (CR) and partial response (PR).
Overall survival (OS) | Baseline up to 96 weeks
  OS defined as the time from the first dose to death from any cause. Survival time was censored at the date of last contact for patients who were still alive or lost to follow-up.
Disease control rate（DCR） | Baseline up to 96 weeks
  Percentage of subjects achieving complete response (CR) and partial response (PR) and stable disease (SD).

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Huashan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer institute and Hospital, Tianjin, Tianjin Municipality